CLINICAL TRIAL: NCT02350725
Title: A Single Center, Randomized, Open-label, Cross-over Exploratory Study to Evaluate the Pharmacodynamic and Pharmacokinetic Response to a Subcutaneous Administration or Oral Administration of Furosemide in Subjects With Heart Failure Presenting With Chronic Fluid Overload
Brief Title: Furosemide Pharmacodynamics and Pharmacokinetics After Subcutaneous or Oral Administration
Acronym: FUROPHARM-HF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: scPharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SCP-01-001; 2014-002546-49 (EudraCT Number)
Record Dates: First submitted 2014-12-09; First posted 2015-01-30 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2014-12

CONDITIONS: Heart Failure
Keywords: Chronic Fluid Overload
MeSH Terms: conditions — Heart Failure | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Furosemide injection solution for subcutaneous administration (80 mg) over 5 hours followed by Oral Furosemide tablets (80 mg) in second period.
  Interventions: Drug: Furosemide injection solution for subcutaneous administration (80 mg); Drug: Oral Furosemide tablets (80 mg)
- Group 2 (Experimental): Oral Furosemide tablets (80 mg) followed by Furosemide injection solution for subcutaneous administration (80 mg) over 5 hours in second period.
  Interventions: Drug: Furosemide injection solution for subcutaneous administration (80 mg); Drug: Oral Furosemide tablets (80 mg)

INTERVENTIONS:
Drug: Furosemide injection solution for subcutaneous administration (80 mg)
Drug: Oral Furosemide tablets (80 mg)

SUMMARY:
The purpose of this pilot study is to investigate the pharmacodynamic and pharmacokinetic parameters of a novel furosemide formulation administered subcutaneously as compared to oral furosemide.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before any assessment is performed
* Male and female subjects ≥18 years of age, with body weight <120 kg and body mass index (BMI) <30 kg/m2
* Female subjects must be at least 2 years post-menopausal
* Participant must have been on oral furosemide (40 mg oid or bid) or therapeutic equivalent (bumetanide 1 mg oid or bid) for a period 90 days before the first dose of study medication
* History of chronic heart failure according to 2012 ESC guidelines with presence of moderate symptoms of chronic fluid overload. Chronic fluid overload is defined as presence of stable signs and symptoms of heart failure and congestion, like dyspnea at mild exertion or minimal exertion, pulmonary congestion and/or peripheral edema at the time of presentation in combination with elevated levels on natriuretic peptides (NT-proBNP > 300 ng/L)
* In the opinion of the investigator, able to participate in the study

Exclusion Criteria:

* Acute Decompensated Heart Failure (ADHF) or recent history of ADHF or significant worsening in their HF symptoms (within prior 2 weeks)
* Contraindication to furosemide
* Systolic BP (SBP) < 90 mm Hg
* Temperature > 38°C (oral or equivalent) or sepsis or active infection requiring i.v. anti-microbial treatment
* Serum sodium < 130 mmol/L and Serum potassium < 3.0 mmol/L
* Current or planned (throughout the completion of study drug infusion) treatment with any i.v. therapies, including inotropic agents, vasopressors, levosimendan, nesiritide or analogues; or mechanical support (intra-aortic balloon pump, endotracheal intubation, mechanical ventilation, or any ventricular assist device)
* History of gastric or intestinal surgery that may affect absorption of oral medication
* Presence or need for urinary catheterization
* Current or planned ultrafiltration, hemofiltration, or dialysis
* Impaired renal function defined as an estimated glomerular filtration rate (eGFR) on admission < 30 mL/min/1.73 m2 will be calculated as per standard at local laboratory
* Administration of intravenous radiographic contrast agent within 72 hours prior to screening or acute contrast-induced nephropathy at the time of screening
* Major surgery within 30 days prior to screening
* Administration of an investigational drug or implantation of investigational device, or participation in another trial, within 30 days before screening
* Inability to follow instructions or comply with procedures
* Any surgical or medical condition which in the opinion of the investigator may interfere with participation in the study or which may affect the outcome of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Diuresis and natriuresis | 8 hours
  Statistical summaries with a graphical presentation will show mean and individual diuresis and natriuresis time profiles such as time to first void, volume of first void, diuresis and natriuresis measured at 60 minute intervals up to 480 minutes following furosemide injection solution for subcutaneous administration or oral tablets. The diuretic response will be compared between therapies using t-tests or Wilcoxon test.

SECONDARY OUTCOMES:
Body Water Content | 8 hours
  The correlation (Pearson coefficient) between bioimpedance (body water content) and diuresis will be investigated including bioimpedance measurement of fluid overload as a predictor diuretic response.
Pharmacokinetic profiles | 8 hours
  A graphical presentation showing mean and individual plasma furosemide concentration-time profiles for comparison between subcutaneous or oral administration. Plasma furosemide concentration-time data will be analyzed using a non-compartmental method and population PK approach (non-linear mixed-effect model). Furosemide concentrations will be summarized using descriptive statistics (including N, mean, standard deviation (SD), coefficient of variation (CV%), median, minimum and maximum) for each treatment.
Cardiac Markers (NTpro-BNP, hs-Trop T, galectin-3) | 8 hours
  Correlation methods to investigate interaction between cardiac makers (NTpro-BNP, hs-Trop T, galectin-3) and pharmacodynamic parameters (diuresis and natriuresis).
Dypsnea Scores on Visual Analog Scale and Likert Scale | 8 hours
  Dyspnea score (Dyspnea Visual Analog Scale and Likert Scale), the New York Heart Association (NYHA) Functional Classification and thirst distress and grading assessments by subjects in response to subcutaneous or oral administration.
Injection site reaction on Draize Scale and Visual Analog Pain Scale | 8 hours
  Visual inspection of injection site, 5-point Draize Scale and Visual Analog pain assessment recorded during subcutaneous administration.

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf A. de Boer, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands